CLINICAL TRIAL: NCT04531904
Title: Prospective Evaluation to Characterize the Real-World Performance of the EMBOVAC Aspiration Catheter for Neurothrombectomy: A Post-Market Clinical Follow-up Trial.
Brief Title: Prospective Evaluation to Characterize the Real-World Performance of the EMBOVAC Aspiration Catheter
Acronym: PERFECT
Status: Completed | Type: Observational
Sponsor: Cerenovus, Part of DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNV_2019_01
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Results first posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-05

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; perfect; embovac
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples Without DNA — Blood Clot / Thrombus
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: EMBOVAC Aspiration Catheter — The EMBOVAC Aspiration catheter is used to treat acute ischemic stroke. The catheter can be used to facilitate introduction of diagnostic or therapeutic agents and is also intended for use in removal/aspiration of emboli and thrombi from selected blood vessels in the neuro vasculature.

SUMMARY:
A post-market study evaluating the EMBOVAC Aspiration Catheter in acute ischemic stroke patients with confirmed intracranial large vessel occlusion.

DETAILED DESCRIPTION:
The PERFECT Study is a prospective, multi-center, single arm, post-market clinical follow-up study.

The objective of this post-market clinical follow-up study is to assess the performance of the EMBOVAC Aspiration Catheter in the treatment of acute ischemic stroke in a real-world clinical setting.

The study will also report on clot characteristics and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥ 18 years old.
2. Subject experiencing acute ischemic stroke with angiographic confirmation of Large Vessel Occlusion of the distal intracranial internal carotid artery, middle cerebral artery or anterior cerebral artery
3. A clinical decision has been made to use the EMBOVAC™ aspiration catheter prior to enrollment in the research
4. EMBOVAC™ Aspiration Catheter is attempted to be used for the first 3 clot removal passes for the target intracranial occlusion
5. Pre-stroke mRS ≤ 1
6. NIHSS ≤ 30
7. Informed Consent has been provided by the subject or the subject's legally authorized representative.

Exclusion Criteria

1. Potential study candidate has already undergone standard of care assessments or treatment that deviate from the clinical research protocol requirements
2. All patients with severe hypertension on presentation. All patients, in whom intravenous therapy with blood pressure medications is indicated, with hypertension that remains severe and sustained despite intravenous antihypertensive therapy
3. Known cerebral vasculitis.
4. Known cancer with life expectancy less than 12 months.
5. Stenosis, or any occlusion, in a vessel proximal to the target occlusion that requires treatment or prevents access to the site of occlusion.
6. Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of recent/ fresh hemorrhage on presentation.
7. Baseline computed tomography (CT) or MRI showing mass effect or intracranial tumor (except small meningioma).
8. Evidence of dissection in the extra or intracranial cerebral arteries.
9. Occlusions in multiple vessels.
10. Confirmation of positive pregnancy test according to site specific standard of care (e.g. test, verbal communication).
11. Currently participating in an investigational clinical trial that may confound study endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Ischemic Stroke patients with confirmed intracranial large vessel occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyriakos Lobotesis, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (2):
- Asklepios Klinik Altona, Hamburg, Germany
- Imperial College Healthcare NHS Trust, London, United Kingdom

REFERENCES:
- [Derived] Piano M, Jansen O, Marnat G, Gory B, Nordmeyer H, Eckert B, Pedicelli A, Cognard C, Loehr C, Zanoni M, Schaefer A, Macera A, Fiehler J, Doyle K, Lobotesis K. Prospective evaluation to characterize the real-world performance of the EMBOVAC aspiration catheter for neurothrombectomy: a post-market clinical follow-up trial. J Neurointerv Surg. 2025 Feb 14;17(3):254-260. doi: 10.1136/jnis-2023-021407. PMID 38609174

RESULTS

PARTICIPANT FLOW:
Groups:
- EMBOVAC Aspiration Catheter: Participants with acute ischemic stroke evaluated by the physician (in accordance with their institutional practice) were attempted with EMBOVAC aspiration catheter or aspiration procedure was performed on Day 0.
Period: Overall Study
Arm/Group | EMBOVAC Aspiration Catheter
Started (Enrolled, attempted and had EmboVAC procedure performed.) | 102
Attempted EmboVac Procedure But Not Performed | 2 (Participants who were not included in the device effectiveness analysis.)
Completed | 87
Not Completed | 15
Not completed — Lost to Follow-up | 1
Not completed — Death | 14

BASELINE CHARACTERISTICS:
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.6 (13.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Revascularization
Description: Successful revascularization was defined as achieving a final modified thrombolysis in cerebral infarction (mTICI) score of 2b or greater in target vessel. Revascularization was measured by an independent adjudicating imaging core laboratory and were reported using expanded treatment in cerebral infarction (eTICI) scale. eTICI was a 7-point grading system for determining response of thrombolytic therapy for ischemic stroke: 0=No reperfusion; 0 percent(%) filling of downstream territory; 1=Thrombus reduction without any reperfusion of distal arteries; 2a=Reperfusion in less than half (1-49%) of the territory; 2b=2b50 (reperfusion in [50-66%] of downstream territory) and 2b67 (reperfusion in (67-89%) of downstream territory); 2c=Reperfusion in [90-99%] of downstream territory; 3=Complete and 100% reperfusion where higher score indicated more successful revascularization.
Time Frame: Day 0 (post-procedure)
Population: The modified intent-to-treat (mITT) analysis set consisted of enrolled participants who received treatment (at least one pass; a pass was defined as use of aspiration followed by evaluation of revascularization with angiography) with the study device. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 99
Percentage of participants | 98.0 [92.9 to 99.8]

2. Secondary Outcome: Percentage of Participants With Successful Revascularization Without Rescue Therapy
Description: Percentage of participants with successful revascularization without rescue therapy was reported. In this outcome measure, successful revascularization was defined as achieving a final mTICI score of 2b or greater in the target vessel as determined by the Independent Imaging Core Laboratory without use of rescue therapy.
Time Frame: Day 0
Population: The mITT analysis set consisted of enrolled participants who received treatment (at least one pass; a pass was defined as use of aspiration followed by evaluation of revascularization with angiography) with the study device. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 99
Percentage of participants | 87.9 [79.8 to 93.6]

3. Secondary Outcome: Percentage of Participants With Complete Revascularization
Description: Complete revascularization was defined as achieving a final mTICI score of 2c or greater in the target vessel as determined by the Independent Imaging Core Laboratory. Revascularization was measured by an independent adjudicating imaging core laboratory and were reported using expanded treatment in cerebral infarction(eTICI) scale. eTICI was a 6-point grading system for determining response of thrombolytic therapy for ischemic stroke:0=No reperfusion; 0 percent (%) filling of downstream territory;1=Thrombus reduction without any reperfusion of distal arteries;2a=Reperfusion in less than half (1-49%) of territory; 2b=2b50 (reperfusion in [50-66%] of downstream territory) and 2b67 (reperfusion in (67-89%) of downstream territory);2c=Reperfusion in [90-99%] of downstream territory;3=Complete and 100% reperfusion where higher score indicated successful revascularization.
Time Frame: Day 0
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 99
Percentage of participants | 86.9 [78.6 to 92.8]

4. Secondary Outcome: Percentage of Participants With First Pass Effect Without Rescue Therapy
Description: Percentage of participants with first pass effect without rescue therapy (mTICI score of 2c or greater after the first pass with the EMBOVAC Aspiration Catheter as determined by the Independent Imaging Core Laboratory) was reported. First pass effect was described as a complete revascularization obtained after a single device pass with no rescue therapy.
Time Frame: Day 0
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 99
Percentage of participants | 53.5 [43.2 to 63.6]

5. Secondary Outcome: Percentage of Participants With Modified First Pass Effect
Description: Percentage of participants with modified first pass effect was reported. Modified first pass effect was defined as mTICI of 2b or greater after the first pass with the EMBOVAC aspiration catheter as determined by the Independent Imaging Core Laboratory.
Time Frame: Day 0
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 99
Percentage of participants | 72.7 [62.9 to 81.2]

6. Secondary Outcome: Time to Recanalization
Description: Time (in minutes) to recanalization (reopening of a previously occluded passageway within a blood vessel) was defined as the procedure time from arterial puncture to recanalization (achievement of the first mTICI score >=2b as determined by the core laboratory) or visualization of final angiographic result if an mTICI score of 2b or greater was not achieved".
Time Frame: Day 0
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 71
Minutes | 27.8 (20.58)

7. Secondary Outcome: Percentage of Participants With Modified Rankin Scale (mRS) Scores 0 to 2 at Day 90
Description: Percentage of participants with mRS scores 0 to 2 at 90 days was reported. The mRS is a scale commonly used to measure the degree of disability or dependence in the daily activities in participants following stroke or other neurological event. It was a 7-point scale that ranged from 0 to 6 where 0=no symptoms at all; 1=no significant disability despite symptoms; 2=slight disability; 3=moderate disability; 4=moderately severe disability; 5=severe disability; 6=death. A lower number indicated lower disability. The mRS evaluation at 90 days was performed by an independent assessor.
Time Frame: at Day 90
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 99
Percentage of participants | 56.6 [46.2 to 66.5]

8. Secondary Outcome: Percentage of Participants With Device Related Serious Adverse Events (SAEs)
Description: SAE was any untoward medical occurrence that at any dose may result in death,life-threatening illness or injury, permanent impairment of body structure or body function including chronic diseases, in-patient or prolonged hospitalization, medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to body structure or body function, fetal distress, fetal death or congenital abnormality or birth defect including physical or mental impairment. Serious adverse device effect was adverse device effect that was resulted in any of consequences characteristic of SAE. Any device related serious adverse event associated with the use of EMBOVAC Aspiration Catheter (or cannot be ruled out as having caused the event) up to 90 days post index stroke procedure. Device relatedness was adjudicated by an independent Clinical Events Committee (CEC).
Time Frame: Up to Day 90 post procedure on Day 0
Population: The safety analysis set consisted of all enrolled participants in whom the procedure was attempted, defined by the advancement of the EMBOVAC Aspiration Catheter inside the participant.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 102
Percentage of participants | 1.0 [0.1 to 6.8]

9. Secondary Outcome: Percentage of Participants With Symptomatic Intracerebral Hemorrhage (sICH)
Description: Percentage of participants with sICH according to Heidelberg Bleeding Classification at 24 hours (hr) post procedure was reported. sICH:new intracranial hemorrhage detected by brain imaging (measured 24 hr post intervention) associated with any of item:>=4 points total National Institute of Health Stroke Scale (NIHSS:tool used by healthcare providers to objectively quantify impairment caused by stroke) at time of diagnosis compared to immediately before worsening; >=2 point in 1 NIHSS category. Rationale:to capture new hemorrhages that produced new neurological symptoms, making it clearly symptomatic but not causing worsening in original stroke territory; lead to intubation/hemicraniectomy/external ventricular drain placement or other major medical/surgical intervention or absence of alternative explanation for deterioration. Independent imaging core laboratory reviewed all 24 hr imaging to identify all ICH. Independent Clinical Events Committee judged ICH as symptomatic/asymptomatic.
Time Frame: 24 hours post procedure on Day 0
Population: The safety analysis set consisted of all enrolled participants in whom the procedure was attempted, defined by the advancement of the EMBOVAC Aspiration Catheter inside of the participant. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 101
Percentage of participants | 0 [0.0 to 3.6]

10. Secondary Outcome: Change From Baseline in National Institutes of Health Stroke Scale (NIHSS) Total Score at 24 Hours Post-procedure
Description: Change from baseline in NIHSS total Score at 24 hours post procedure was reported. NIHSS is an assessment which objectively quantifies the impairment caused by stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, 0=normal function in that specific ability, while a higher score (4)=some level of impairment. The individual scores from each item are summed in order to calculate a participant's total NIHSS score. The participant's total NIHSS score ranges from 0 (minimum) - 42 (maximum). Score 0 (no stroke symptoms); 1 - 4 (Minor stroke); 5-15 (Moderate stroke); 16-20 (Moderate to severe stroke); and 21-42 (Severe stroke).
Time Frame: Baseline (Day 0, before procedure) up to 24 hours post procedure on Day 0
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 101
Scores on a scale | -6.9 (6.36)

11. Secondary Outcome: Number of Participants With All-Cause Mortality Thorugh 90 Days
Description: Number of participants with all-cause mortality through 90 days post procedure was reported. All-cause mortality included all deaths of participants due to any cause. Participants without events were censored at the date of last contact in the study.
Time Frame: 90 days post procedure on Day 0
Population: The safety analysis set consisted of all enrolled participants in whom the procedure was attempted, defined by the advancement of the EMBOVAC Aspiration Catheter inside of the participant.
Measure: Count of Participants; unit: Participants
Arm/Group | EMBOVAC Aspiration Catheter
Number analyzed (Participants) | 102
Participants | 13

ADVERSE EVENTS:
Time Frame: Serious adverse events and Other adverse events (Non-serious): Up to Day 90; for all-cause mortality: From Day 0 to end of the study (i.e., up to 21.3 months )
Description: The safety analysis set consist of all enrolled participants in whom the treatment was attempted, defined by the advancement of the EMBOVAC Aspiration Catheter inside the participant.
Arm/Group | EMBOVAC Aspiration Catheter
All-Cause Mortality (participants affected / at risk) | 14/102
Serious Adverse Events (participants affected / at risk) | 26/102
Other Adverse Events (participants affected / at risk) | 17/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMBOVAC Aspiration Catheter (N=102)
Cerebral artery occlusion (Nervous system disorders) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 2 (2)
Haemorrhagic transformation stroke (Nervous system disorders) | 2 (2)
Brain oedema (Nervous system disorders) | 1 (1)
Stroke in evolution (Nervous system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 2 (2)
Endocarditis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrioventricular block (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intraoperative cerebral artery occlusion (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site occlusion (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMBOVAC Aspiration Catheter (N=102)
Haemorrhagic transformation stroke (Nervous system disorders) | 9 (9)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2)
Cerebral artery perforation (Nervous system disorders) | 1 (1)
Cerebral microhaemorrhage (Nervous system disorders) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Air embolism (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 2 (2)
Organic brain syndrome (Psychiatric disorders) | 1 (1)
Vasospasm (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Draft abstracts, manuscripts, and materials for presentation at scientific meetings must be sent to the sponsor at least 60 working days prior to abstract or other relevant submission deadlines. Authorship of publications resulting from this study was based on generally accepted criteria for major medical journals.

DOCUMENTS (2):
  • Study Protocol (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT04531904/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/04/NCT04531904/SAP_001.pdf